**Document Type:** Informed Consent Form

Official Title: Train Your Brain – Executive Function

NCT Number: NCT05938894

IRB Approval Date: 03/03/2023

**Note:** A stamped consent was provided with the initial IRB protocol approval. Since the study was conducted online and consent was obtained through Qualtrics, a stamped consent was not provided with later IRB approval notices.

# GRAND FORKS HUMAN NUTRITION RESEARCH CENTER CONSENT TO PARTICIPATE IN RESEARCH

Project Title: Train Your Brain

Principal Investigators: James Roemmich, PhD

Julie Hess, PhD

Shanon Casperson, PhD, DTR

**Phone/Email Addresses:** 701-795-8272/James.Roemmich@usda.gov

701-795-8146/Julie.Hess@usda.gov

701-795-8497/Shanon.Casperson@usda.gov

#### What should I know about this research?

• Someone will explain this research to you.

- Taking part in this research is voluntary. Whether you take part is up to you.
- If you don't take part, it won't be held against you.
- You can take part now and later drop out, and it won't be held against you
- If there is anything in this form that you don't understand, ask questions.
- Ask all the questions you want before you decide.

# How long will I be in this research?

We expect that your taking part in this research will last about 10 weeks.

#### Why is this research being done?

The purpose of this research is to test if playing games designed to improve your executive function can change your views about the types of foods you eat. Executive function is a set of mental processes that you use every day to make decisions – such as what kinds of foods you choose to eat and when and where you eat those foods.

# What happens to me if I agree to take part in this research?

If you decide to take part in this research study, you will fill out some questionnaires and do some tasks on a desktop or laptop computer or tablet.

You will fill out some questionnaires at the beginning of the study asking about yourself, your health, your diet and eating behaviors, and your stress. Then 2 hours after you have eaten you will tell us how much you like certain foods and how much you are willing to pay for those foods. For this task a picture of a food will appear on your screen. Below the picture will be a slider that you will use to tell how much you like that food. You will move the slider button to the value that best matches how much you like the food. When happy with your choice you will press submit. After you tell us how much you like that food another slider will appear for you to

Approval Date: \_\_3/3/2023 \_\_\_\_\_

Expiration Date: \_3/2/2024 \_\_\_\_\_

University of North Dakota IRB

tell us how much you would pay for that food. You will move the slider button to the point on the value that best matches how much you would pay for the food. When happy with your choice you will press submit. You will do this for 36 different foods. You will also play 4 games to test your executive function.

# The 4 games are:

- 1. The "Go No-Go" game. For this game pictures will appear on your screen with a solid or dashed line around them. You will only click on the picture when you see a solid line around it. It will take about 10 minutes to play this game.
- 2. The "Dot Probe" game. For this game you will see 2 pictures on your screen for a couple of seconds and then they will go away, and a black dot will appear. You will click on the black dot. The black dot will be in different places on your screen after each set of pictures. It will take about 14 minutes to play this game.
- 3. The "Visual Search" game. For this game you will see 16 pictures on your screen. You will have to find the picture described in the instructions. It will take about 6 minutes to play this game.
- 4. The "Stop Signal" game. For this game pictures will appear on your screen with a red or green line around it. You will only click on the picture when you see a green line around it. It will take about 8 minutes to play this game.

You will play each of these games 2 times each week for 8 weeks. You can play the games as much as you want but you have to play each game at least 2 times every week. You can play the games on your desktop or laptop computer, tablet, or smartphone as long as it has internet access. You do not have to use the same device every time you play games. We will monitor your game play and will send reminders via email or text message if we see that you have not played each game at least 2 times that week.

At the end of 8 weeks, you will fill out some of the same questionnaires about your diet, eating behaviors and stress that you filled out at the beginning of the study. You will also complete the same computer task. You will tell us again how much you like and will pay for certain foods. This will be done 2 hours after you have eaten. You will also play each of the 4 games as you did at the beginning of the study. You will have to play these 4 games on the same desktop or laptop computer, smartphone, or tablet that you did at the beginning of the study.

#### Could being in this research hurt me?

Risks are similar to those encountered in daily life and are considered minimal. However, with any internet use there is a risk of data breach. This risk is minimized by using secure sites for data collection. Also, you do not have to answer any question on the questionnaires that cause you distress.

Approval Date: \_\_3/3/2023 \_\_\_\_\_

Expiration Date: \_3/2/2024 \_\_\_\_\_

University of North Dakota IRB

## Will being in this research benefit me?

It is not expected that you will personally benefit from this research. Possible benefits to others include a simple, inexpensive, readily available tool to help improve a person's executive function.

## How many people will participate in this research?

Approximately 500 people will take part in this study.

## Will it cost me money to take part in this research?

You will not have any costs for being in this research study. But you must have access to the internet. You also need a desktop or laptop computer, smartphone, or tablet on which to complete all the task required by this study. Also, we do not withhold income, social security, unemployment taxes, or any other taxes. You may have to pay income taxes on the money you receive. All tax questions relating to the taxability of the payment should be directed to your personal tax accountant or to your local Internal Revenue Service Office.

# Will I be paid for taking part in this research?

You will be paid for being in this research study. After you finish the study, we will send you a check for \$340. To get this payment you must complete all the tasks mentioned in this form.

## Who is funding this research?

The United States Department of Agriculture (USDA) is funding this research study. This means that the Grand Forks Human Nutrition Research Center is receiving payments from the USDA to support the activities that are required to conduct the study. No one on the research team will receive a direct payment or an increase in salary from the USDA for conducting this study.

## What happens to information collected for this research?

Your private information may be shared with individuals and organizations that conduct or watch over this research, including:

- The USDA, as specified in the USDA/ARS Privacy Act System of Records
- Study personnel who work at the Grand Forks Human Nutrition Research Center
- The Institutional Review Board (IRB) that reviewed this research

We may publish the results of this research. However, we will keep your name and other identifying information confidential. We protect your information from disclosure to others to the extent required by law. We cannot promise complete secrecy. Data collected in this research might be de-identified and used for future research or distributed to another investigator for future research without your consent.

| Approval Date:3/3/2023 |
|--------------------------------|
| Expiration Date: _3/2/2024 |
| University of North Dakota IRB |

# What if I agree to be in the research and then change my mind?

If you decide to leave the study early, we ask that you contact us to let us know. You can contact us by email or by calling any of the numbers listed at the top of this form.

## Who can answer my questions about this research?

If you have questions, concerns, or complaints, or think this research has hurt you or made you sick, talk to the research team at the phone number listed above on the first page.

This research is being overseen by an Institutional Review Board ("IRB"). An IRB is a group of people who perform independent review of research studies. You may talk to them at 701.777.4279 or UND.irb@UND.edu if:

- You have questions, concerns, or complaints that are not being answered by the research team.
- You are not getting answers from the research team.
- You cannot reach the research team.
- You want to talk to someone else about the research.
- You have questions about your rights as a research subject.
- You may also visit the UND IRB website for more information about being a research subject: http://und.edu/research/resources/human-subjects/research-participants.html

By clicking the box below, I certify that:

- I am 18 years old or older.
- I am a U.S. citizen.
- I have read and agree to the terms above.
- I freely consent to participate in this study.

| Checking this box indicates that you are at least 18 years old and a U.S. citizen, you have read and agree to the terms above and you freely consent to participate in this study. |
|---|
| *Please enter your first and last name in the box below: |
| *Please enter your email in the box below: |

| Approval Date: <u>3/3/2023</u> |
|--------------------------------|
| Expiration Date: _3/2/2024 |
| University of North Dakota IRB |